CLINICAL TRIAL: NCT02432287
Title: Metformin in Longevity Study (MILES).
Acronym: MILES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2014-3444
Record Dates: First submitted 2015-02-24; First posted 2015-05-04 (Estimated); Results first posted 2018-05-31 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Aging
Keywords: aging; metformin; prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Metformin, an FDA approved first-line drug for the treatment of type 2 diabetes, has known beneficial effects on glucose metabolism.
  Interventions: Drug: Metformin
- Placebo (Experimental): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — To determine if treatment with metformin (1700 mg/day) will restore the gene expression profile of older, glucose intolerant adults to that of young healthy subjects.
  Other Names: Glucophage
  Arms: Metformin
Drug: Placebo — there is no other name we used for the placebo
  Other Names: no others
  Arms: Placebo

SUMMARY:
Metformin, an FDA approved first-line drug for the treatment of type 2 diabetes, has known beneficial effects on glucose metabolism. Evidence from animal models and in vitro studies suggest that in addition to its effects on glucose metabolism, metformin may influence metabolic and cellular processes associated with the development of age-related conditions, such as inflammation, oxidative damage, diminished autophagy, cell senescence and apoptosis. As such, metformin is of particular interest in clinical translational research in aging since it may influence fundamental aging factors that underlie multiple age-related conditions. The investigators therefore propose a pilot study to examine the effect of metformin treatment on the biology of aging in humans. Namely, whether treatment with metformin will restore the gene expression profile of older adults with impaired glucose tolerance (IGT) to that of young healthy subjects.

DETAILED DESCRIPTION:
Aging in humans is a well-established primary risk factor for many disabling diseases and conditions, among them diabetes, cardiovascular disease, Alzheimer's disease and cancer. In fact, the risk of death from these causes is dramatically accelerated (100-1000 fold) between the ages of 35 and 85 years. For this reason, there is a need for the development of new interventions to improve and maintain health into old age - to improve "healthspan".

Several mechanisms have been shown to delay the aging process, resulting in improved healthspan in animal models, including mammals. These include caloric restriction, alteration in GH/IGF1 pathways, as well as use of several drugs such as resveratrol (SIRT1 activator) and rapamycin (mTOR inhibitor). At Einstein, the investigators have been working to discover pathways associated with exceptional longevity. The investigators propose the study of drugs already in common clinical use (and FDA approved) for a possible alternative purpose -healthy aging. The investigators goal is to identify additional mechanisms involved in aging, the delay of aging and the prevention of age-related diseases. In this proposal, the investigators explore the possibility of a commonly used drug, metformin, to reverse relevant aspects of the physiology and biology of aging.

Metformin is an FDA approved drug in common use in the US since the 1990s. It is the first-line drug of choice for prevention and treatment of type 2 diabetes (T2DM). The effect of metformin on aging has been extensively studied, and has been associated with longevity in many rodent models. Metformin also extends the lifespan of nematodes, suggesting an evolutionarily conserved mechanism. A recent high impact study demonstrated that metformin reduces oxidative stress and inflammation and extends both lifespan and health span in a mouse model .

If indeed metformin is an "anti-aging" drug, its administration should be associated with less age-related disease in general, rather than the decreased incidence of a single age-related disease. This notion led investigators to further study whether anti-aging effects can be demonstrated in the type 2 diabetes population. Notably, in the United Kingdom Prospective Diabetes Study (UKPDS) metformin, compared with other anti-diabetes drugs, demonstrated a decreased risk of cardiovascular disease. This has been suggested in other studies and meta-analyses and remains an active area of research.

In addition, numerous epidemiologic studies have shown an association of metformin use with a decreased risk of cancer, as well as decreased cancer mortality. There is also evidence from studies performed both in-vitro and in-vivo of metformin's role in attenuating tumorigenesis. The mechanisms proposed relate to its effects on reducing insulin levels, improved insulin action, decreased IGF-1 signaling (central to mammalian longevity), as well as activation of AMP-kinase. In fact, metformin's potential protective effect against cancer has been gaining much attention, with over 100 ongoing studies registered on the Clinical Trials.gov website.

To characterize pathways associated with increased lifespan and healthspan, the investigators plan to compile a repository of muscle and adipose biopsy samples obtained from young healthy subjects and older adults before and after treatment with potential anti-aging drugs. RNA-Seq analysis will be used to identify a unique biological "fingerprint" for aging in these tissues by comparing changes in gene expression in older adults post-drug therapy to the profiles of young healthy subjects. This overall approach is supported by a grant from the Glenn Foundation for the Study of the Biology of Human Aging.

The investigators believe that if metformin changes the biology of aging in tissues to a younger profile, it supports the notion that this drug may have more widespread use - as an "anti-aging" drug.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women;
2. age >60 years with IGT based on 75g OGTT (fasting plasma glucose < 126 mg/dl, 2-hr glucose between 140 - 199 mg/dl);
3. this definition of IGT will include individuals with combined impaired fasting glucose (IFG) and IGT.

The investigators chose these inclusion criteria in order to study subjects who have evidence of impaired glucose regulation, but are not yet diabetic.

Exclusion Criteria:

1. Serious chronic or acute illness: cancer, clinically significant congestive heart failure, COPD, inflammatory conditions, serum creatinine > 1.4 mg/dl (female) or > 1.5 mg/dl (male), active liver disease, history of metabolic acidosis, poorly controlled hypertension, epilepsy, recent (within 3 months) CVD event (MI, PTCA, CABG, stroke); history of bariatric or other gastric surgery, cigarette smoking, binge alcohol use (>7 drinks in 24 hrs).
2. Treatment with drugs known to influence glucose metabolism (other diabetes medications, systemic glucocorticoids, pharmacologic doses of niacin)
3. Hypersensitivity to metformin or any component of the formulation

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Crandall, MD, Principal Investigator — Einstein College of Medicine
Locations (1):
- Einstein College of Medicine of Yeshiva University, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin First, Then Placebo: Metformin, an FDA approved first-line drug for the treatment of type 2 diabetes, has known beneficial effects on glucose metabolism.
  Participants in the metformin first group took 1-2 metformin capsules 2 times daily for 6 weeks, followed by a 2 week washout period, concluding with 6 weeks of 1-2 placebo capsules (which matched metformin capsules) 2 x daily.
- Placebo First, Then Metformin: Participants in the placebo first group took 1-2 placebo capsules 2 x daily (which matched metformin capsules) for 6 weeks, followed by a 2 week washout period, concluding with 6 weeks of 1-2 metformin capsules 2x daily.
Period: First Intervention
Arm/Group | Metformin First, Then Placebo | Placebo First, Then Metformin
Started | 8 | 8
Completed | 8 | 7
Not Completed | 0 | 1
Period: Washout Period
Arm/Group | Metformin First, Then Placebo | Placebo First, Then Metformin
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Metformin First, Then Placebo | Placebo First, Then Metformin
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Metformin FIRST, Then Placebo: Metformin, an FDA approved first-line drug for the treatment of type 2 diabetes, has known beneficial effects on glucose metabolism.
  In the metformin first group, individuals took 1700mg/day metformin in 2 doses for 6 weeks, followed by 2 weeks of washout, and concluding with placebo capsules that matched the metformin for 6 weeks.
- Placebo FIRST, Then Metformin: In the placebo first group, individuals took placebo capsules that matched metformin for 6 weeks, followed by 2 weeks of washout, and concluding with metformin 1700mg/day (in 2 doses) for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Metformin FIRST, Then Placebo | Placebo FIRST, Then Metformin | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (6.7) | 74 (5.4) | 71 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28 (3.1) | 32 (4.4) | 30 (4.3)
Weight [Mean (Standard Deviation); unit: kg] | 84 (14) | 89 (17) | 87 (16)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 108 (13) | 102 (10) | 105 (12)
2-hour glucose [Mean (Standard Deviation); unit: mg/dL] | 153 (13) | 171 (24) | 162 (21)
Antihypertensive therapy [Count of Participants; unit: Participants] | 5 | 6 | 11
Statin therapy [Count of Participants; unit: Participants] | 3 | 3 | 6
Aspirin therapy [Count of Participants; unit: Participants] | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Increase in Number of Expressed Genes in Muscle and Adipose Tissue Using RNA Sequencing (RNA-Seq)
Description: The investigators hypothesize that treatment with metformin will result in changes in the transcriptome. The investigators will test this by identifying increases in gene expression in muscle and adipose tissue with RNA Sequencing (RNA-Seq) in metformin and in placebo.
Time Frame: 6 weeks
Measure: Number; unit: genes
Groups:
- Metformin Treatment: Metformin, an FDA approved first-line drug for the treatment of type 2 diabetes, has known beneficial effects on glucose metabolism.
  Participants took metformin (1700 mg/day) for 6 weeks, followed by a 2 week washout, concluding with placebo pills (that matched metformin) for 6 weeks.
- Placebo Treatment: Participants took placebo that matched metformin for 6 weeks.
Arm/Group | Metformin Treatment | Placebo Treatment
Number analyzed (Participants) | 14 | 14
genes
  genes increased in muscle | 245 | 402
  genes increased in adipose | 15 | 132

2. Secondary Outcome: Mixed Meal Tolerance. Assessment of Insulin Sensitivity and Insulin Secretion (Using a Modification of the Matsuda Index)
Description: Assessment of insulin sensitivity and insulin secretion. Insulin sensitivity will be estimated from insulin and glucose levels obtained following the standard meal challenge, using a modification of the Matsuda index, which has been widely used for non-invasive assessment of insulin sensitivity and shows good correlation (r=0.73) with results obtained from euglycemic hyperinsulinemic clamp studies. A higher Matsuda index indicates better insulin sensitivity. The insulin sensitivity index (ISI (comp) was calculated using the following equation (where g denotes glucose at various time points and i denotes insulin at various time points): ISI (comp)= 10000/ ((g0*i0* ((g0*15+ g30*30+ g60*30+ g90*30+ g120*30+ g180*30+ g240*15)/240))* ((i0*15+ i30*30+ i60*30+ i90*30*+ i120*30+ i180*30+ i240*15)/240))^0.5
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: index
Groups:
- Metformin Treatment: Metformin, an FDA approved first-line drug for the treatment of type 2 diabetes, has known beneficial effects on glucose metabolism.
  During metformin treatment, individuals took 1700mg/day metformin in 2 doses for 6 weeks.
- Placebo Treatment: During the placebo treatment, individuals took placebo capsules that matched metformin for 6 weeks.
Arm/Group | Metformin Treatment | Placebo Treatment
Number analyzed (Participants) | 14 | 14
index | 5.6 (3.9) | 4.1 (2.1)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the study period of 14 weeks.
Groups:
- Metformin: Metformin, an FDA approved first-line drug for the treatment of type 2 diabetes, has known beneficial effects on glucose metabolism.
  Participants took metformin capsules 2 times daily for 6 weeks.
- Placebo: All participants took placebo capsules 2 x daily for 6 weeks.
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=15) | Placebo (N=15)
Hematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Hematoma of thigh after muscle biopsy.
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant developed nausea and vomiting after taking opiate analgesic for hematoma
urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) — Participant developed urinary retention during study treatment requiring foley catheter placement.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=15) | Placebo (N=15)
Shingles (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Participant developed shingles during study
Chest pain (Cardiac disorders) | 0 (0) | 1 (1) — Participant developed an episode of 4 minutes of chest pain and palpitations during study treatment.

LIMITATIONS AND CAVEATS:
Limitations:

Crossover design may lead to a carryover effect that was not detected due to small sample size.

The sample size was small and certain genes that were differentially expressed may not have been detected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No